CLINICAL TRIAL: NCT02439580
Title: Effect of Annona Muricata Leaves on Nutritional Status, Quality of Life, Fecal Butyrate, Inflammation, and Colorectal Cancer Cells
Brief Title: Effect of Annona Muricata Leaves on Colorectal Cancer Patients and Colorectal Cancer Cells
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Lili Indrawati, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 406/H2.F1/ETIK/2013
Record Dates: First submitted 2015-04-27; First posted 2015-05-12 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Colorectal Cancer
Keywords: Patients; After Surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Annona muricata extract (Experimental): Annona muricata ethanol-soluble fraction of water extract capsule, 300 mg/day, for eight weeks
  Interventions: Dietary Supplement: Annona muricata extract
- Placebo (Placebo Comparator): Maltose capsule, 300 mg/day, for eight weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Annona muricata extract — ethanol-soluble fraction of water extract
  Arms: Annona muricata extract
Dietary Supplement: Placebo — maltose
  Arms: Placebo

SUMMARY:
Annona muricata L., include the leaves, is found to contain biologically active Annonaceous acetogenins and plant polyphenols that are important components of human diet and a number of them are considered to have chemopreventive and therapeutic properties against cancer.

To confirm previous findings in in vitro, animal study and traditionally use, a human, ex vivo and in vitro studies were conducted to evaluate the effects of consecutive ingestion of A. muricata leaves extract for eight weeks.

DETAILED DESCRIPTION:
Colorectal cancer patients were randomly assigned to receive either A. muricata leaves extract or placebo. Dietary intakes and anthropometry were assessed with food record every two weeks. Blood parameters, nutritional status, quality of life, fecal butyrate level, and systemic inflammation of patient were assessed at the beginning and the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Colorectal Carcinoma
* Have undergone standard therapy
* Satisfactory haematological or biochemical functions
* Karnofsky performance status of ≥ 60%
* Willing not to take probiotic supplement during study period

Exclusion Criteria:

* Uncontrolled hypertension
* Serious heart, kidney, liver endocrine or neurologic/psychiatric diseases
* Physical and mental disability that renders them unable to verbally communicate
* History of recent cancers
* Pregnant, lactating, or not using adequate contraception
* Patient on other investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Nutritional Status | eight weeks

SECONDARY OUTCOMES:
Cytotoxicity | two days
  Cytotoxicity against colorectal cancer cell lines that were treated with serum of participants, is assessed by MTT assay

CONTACTS AND LOCATIONS:
Overall Officials: Lili Indrawati, MSc, Principal Investigator — Indonesia University